CLINICAL TRIAL: NCT01120366
Title: Success of Tocilizumab in RA Patients With Remission Induction and Sustained Efficacy After Discontinuation
Acronym: SURPRISE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: SURPRISE Study Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SURPRISE Study; UMIN000002744 (Other: UMIN)
Record Dates: First submitted 2010-05-06; First posted 2010-05-10 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SWITCH (Active Comparator): Tocilizumab monotherapy
  Interventions: Drug: Tocilizumab
- ADD-ON (Active Comparator): Tocilizumab plus methotrexate combination
  Interventions: Drug: Tocilizumab plus methotrexate

INTERVENTIONS:
Drug: Tocilizumab plus methotrexate — Tocilizumab 8mg/kg 4weeks (i.v.) plus methotrexate up to 52weeks.The dosage of MTX will be fixed at least 24 weeks from the start of the study.
  Other Names: Actemra; Methotrexate
  Arms: ADD-ON
Drug: Tocilizumab — tocilizumab 8mg/kg/4weeks (i.v.) up to 52weeks.
  Other Names: Actemra
  Arms: SWITCH

SUMMARY:
The objective of this study is to investigate the efficacy and safety of the humanized anti-human IL-6 receptor monoclonal antibody tocilizumab (TCZ) either in monotherapy or in combination therapy with methotrexate (MTX) in patients with an inadequate response to treatment with MTX.

Furthermore, in patients who have been able to achieve control of disease activity via the above therapy, we investigate the possibility of stopping TCZ and verify safety when TCZ is restarted after disease recurrence.

DETAILED DESCRIPTION:
In this study, we aim to prospectively and randomly evaluate efficacy for changes in clinical remission and joint destruction in RA patients in treatment with TCZ monotherapy(SWITCH) and in combination therapy with MTX(ADD-ON), and also to investigate the best therapeutic approach to achieve discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with RA in accordance with the 1987 classification criteria of ACR
* Aged 20 to 75 years inclusive at enrolment (within 2 weeks before starting treatment with the investigational drug)
* Treated with MTX at ≥6 mg/week for at least 8 weeks immediately before enrolment
* Rheumatoid arthritis of duration ≤10 years
* DAS28-ESR ≥3.2 (within 2 weeks before starting treatment with the investigational drug)
* Having received and thoroughly understood an adequate explanation about participation in the study, patients who have personally and voluntarily provided written informed consent

Major exclusion criteria:

* Patients who were Steinbrocker Class IV.
* Patients who received leflunomide within 12 weeks, DMARDs other than MTX within 8 weeks , or tacrolimus within 4 weeks before the 1st TCZ infusion.
* Patients who previously received biologic DMARDs including TCZ.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2009-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
DAS28-ESR remission at 24 weeks | at 24 week
  Step 1: Investigation of the efficacy and safety of TCZ in combination therapy with MTX
Changes over time in the number of patients maintaining discontinuation (maintenance rate) | Week 52 to Week 104
  Step 2: Investigation of discontinuation

SECONDARY OUTCOMES:
Change in TSS score | at 52 weeks (after treatment initiation)
  Step 1
Change of DAS28-ESR remission rate | Week 0 to Week 52
  Step 1
Change of ACR response rate | Week 0 to Week 52
  Step 1
EQ5D scores over time | Week 0 to Week 52
  Step 1
J-HAQ/HAQ scores over time | Week 0 to Week 52
  Step 1
SDAI, CDAI, and Boolean remission rates | Week 0 to Week 52
  Step 1
TNF-α over time | Week 0 to Week 52
  Step 1
Between-group comparison of the discontinuation rate after an achievement of remission | Week 0 to Week 104
  Step 2
Factor analysis of patients maintaining discontinuation | Week 0 to Week 104
  Step 2
Time course of DAS28 after restarting TCZ (between-group comparison) | Week 52 to Week 104
  Step 2
Change in TSS score | Week 52 to Week 104
  Step 2
Time course of DAS28 after restarting MTX following suspension of discontinuation in the TCZ monotherapy group in Step 1 | Week 52 to Week 104
  Step 2
SDAI, CDAI, and Boolean remission rates | Week 52 to Week 104

OTHER OUTCOMES:
Adverse events | During the study period

CONTACTS AND LOCATIONS:
Overall Officials: Tsutomu Takeuchi, Principal Investigator — Keio University
Locations (30):
- Japan (30):
  - Hokkaido Medical Center for Rheumatic Diseases Hospital, Sapporo, Hokkaido
  - Utazu Hama Clinic, Ayautagun
  - Graduate School of Medical and Dental Sciences, Tokyo Medical and Dental University, Bunkyō City
  - Fukushima Red-Cross Hospital, Fukushima
  - Higashihiroshima Memorial Hospital, Higashihiroshima
  - Tokyo Dental College Ichikawa General Hospital, Ichikawa
  - Itabashi Medical Center, Itabashi-ku
  - Shimane University Faculty of Medicine, Izumo
  - Saitama Medical Center, Saitama Medical University, Kawagoe
  - Kagawa University, Kida-gun
  - University of Occupational and Environmental Health Hospital, Kitakyushu
  - Kurashiki Sweet Hospital, Kurashiki
  - Kyoto University Graduate School of Medicine, Kyoto
  - Marunouchi Hospital, Matsumoto
  - Dogo Spa Hospital, Matsuyama
  - Zenjinkai Shimin-no-mori Hospital, Miyazaki
  - Nagasaki University Graduate School of Biomedical Sciences, Nagasaki
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - Niigata University Graduate School of Medical and Dental Sciences, Niigata
  - Department of Internal Medicine, Hyogo College of Medicine, Nishinomiya
  - Oribe Rheumatism and Internal Medicine Clinic, Ōita
  - Hokkaido University Graduate School of Medicine, Sapporo
  - Sasebo Chuo Hospital, Sasebo
  - Niigata Rheumatic Center, Shibata
  - Osaka University Hospital, Suita
  - Institute of Rheumatology, Tokyo Women's Medical University, Tokyo
  - Keio University Hospital, Tokyo
  - The University of Tokyo Graduate School of Medicine, Tokyo
  - Tomishiro Chuo Hospital, Tomishiro
  - Yokohama Minami Kyousai Hospital, Yokohama

REFERENCES:
- [Derived] Kato M, Kaneko Y, Tanaka Y, Inoo M, Kobayashi-Haraoka H, Amano K, Miyata M, Murakawa Y, Yasuoka H, Hirata S, Nagasawa H, Tanaka E, Miyasaka N, Yamanaka H, Yamamoto K, Yokota I, Atsumi T, Takeuchi T. Predictive value of serum amyloid a levels for requirement of concomitant methotrexate in tocilizumab initiation: A post hoc analysis of the SURPRISE study. Mod Rheumatol. 2020 May;30(3):442-449. doi: 10.1080/14397595.2019.1621026. Epub 2019 Jun 7. PMID 31106666
- [Derived] Kaneko Y, Kato M, Tanaka Y, Inoo M, Kobayashi-Haraoka H, Amano K, Miyata M, Murakawa Y, Yasuoka H, Hirata S, Tanaka E, Miyasaka N, Yamanaka H, Yamamoto K, Takeuchi T; SURPRISE study group. Tocilizumab discontinuation after attaining remission in patients with rheumatoid arthritis who were treated with tocilizumab alone or in combination with methotrexate: results from a prospective randomised controlled study (the second year of the SURPRISE study). Ann Rheum Dis. 2018 Sep;77(9):1268-1275. doi: 10.1136/annrheumdis-2018-213416. Epub 2018 May 31. PMID 29853455
- [Derived] Kaneko Y, Atsumi T, Tanaka Y, Inoo M, Kobayashi-Haraoka H, Amano K, Miyata M, Murakawa Y, Yasuoka H, Hirata S, Nagasawa H, Tanaka E, Miyasaka N, Yamanaka H, Yamamoto K, Takeuchi T. Comparison of adding tocilizumab to methotrexate with switching to tocilizumab in patients with rheumatoid arthritis with inadequate response to methotrexate: 52-week results from a prospective, randomised, controlled study (SURPRISE study). Ann Rheum Dis. 2016 Nov;75(11):1917-1923. doi: 10.1136/annrheumdis-2015-208426. Epub 2016 Jan 5. PMID 26733110